CLINICAL TRIAL: NCT04954118
Title: Use of Aerosol Box for Ultrasound-guided Internal Jugular Vein Cannulation in COVID-19 Patients; Single Center Experience
Brief Title: A Different Use of The Aerosol Box in COVID-19 Patients; Internal Jugular Vein Cannulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Gokhan Sertcakacilar, MD, Principal investigator, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2020-287
Record Dates: First submitted 2021-07-04; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: COVID-19 Pneumonia
Keywords: Aerosol box; SARS-CoV-2 virus; COVID-19; Internal jugular vein; Personal protective equipment
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group P (Active Comparator): The clinicians performed an internal jugular vein cannulation using only personal protective equipment.
  Interventions: Procedure: Internal jugular vein cannulation
- Group P&A (Active Comparator): The clinicians performed an internal jugular vein cannulation using personal protective equipment and aerosol box.
  Interventions: Procedure: Internal jugular vein cannulation

INTERVENTIONS:
Procedure: Internal jugular vein cannulation — The clinicians performed an internal jugular vein cannulation using personal protective equipment (PPE) or both of the aerosol box and PPE provide insertion of a central venous catheter in COVID-19 patients.

SUMMARY:
During the COVID-19 pandemic, health employees are at high risk of infection. This study aimed to determine experiences with an aerosol box (AB), used with the aim of preventing contamination by droplets during internal jugular vein cannulation which requires close contact with COVID-19 patients, and the necessity to use this device.

DETAILED DESCRIPTION:
The study included 40 patients with diagnosis of COVID-19 requiring central venous catheter during treatment in the ward. The patients were randomly allocated to one of the two protective equipment groups and, then, randomly assigned to one of the five clinicians. Group P&A had both personal protective equipment (PPE) and AB used, while Group P included patients where PPE was used alone. Clinicians completed a survey after performing the procedure to evaluate the use of the aerosol box. Collected data of the procedures and patients, were analyzed. In addition, survey data were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with COVID-19 and inserted central venous catheter while being treated in the ward

Exclusion Criteria:

* Patients under the age of 18 years
* Patients who can not lie in the supine position due to severe respiratory distress,
* Patients with thrombus in the right İJV in evaluation with US

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-03-20 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Questionnaire on the Use of Aerosol Boxes | 7 months from the index case of the pandemic in Turkey
  There is no valid and reliable questionnaire in the literature that evaluates behaviors and attitudes towards aerosol box use. Therefore, in our study, a questionnaire was conducted about the attitudes and behaviors of the participants towards aerosol box preservatives.There are 6 statements in the content of the questionnaire on aerosol box use. The questionnaire consists of expressions such as "1-Discomfort using box, 2-Difficulty in manipulation during the performance, 3-Difficulty in use of US device restricted by box, 4-Increased cognitive load from use of box, 5-Increased physical load from use of box, 6-User satisfaction respectively. Participants were asked to answer these statements as ''yes or no''. According to the response received, positive or negative attitudes towards the use of aerosol boxes were evaluated.
Catheter-related infection after central venouse catheterization in COVID-19 | 7 months from the index case of the pandemic in Turkey
  When the body temperature of the patients is above 38, blood, urine and if the patient is intubated, a tracheal aspirate culture will be taken.
  If the blood culture test is a positive, a diagnosis of catheter-related infection will be made and central venouse catheter will be removed.

SECONDARY OUTCOMES:
Number of arterial punctures | 7 months from the index case of the pandemic in Turkey
  The difference in the number of arterial punctures developed during central venous catheterization in patients with or without aerosol box.

CONTACTS AND LOCATIONS:
Locations (1):
- Bakirkoy Dr. Sadi Konuk Research and Training Hospital, Istanbul, Bakirkoy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No